CLINICAL TRIAL: NCT00062751
Title: A Phase 2 Randomized Open-Label Study Of Letrozole In Combination With Two Dose Levels And Schedules Of Oral Temsirolimus (CCI-779), Or Letrozole Alone, In Postmenopausal Women With Locally Advanced Or Metastatic Breast Cancer
Brief Title: Study Evaluating Temsirolimus (CCI-779) In Breast Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3066A1-204; B1771005; NCT00061971 (obsolete NCT alias)
Record Dates: First submitted 2003-06-12; First posted 2003-06-13 (Estimated); Results first posted 2010-11-25 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Breast Neoplasms
Keywords: breast; neoplasms
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Letrozole; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: Letrozole / Temsirolimus (CCI-779)
- B (Experimental)
  Interventions: Drug: Letrozole / Temsirolimus (CCI-779)
- C (Active Comparator)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole / Temsirolimus (CCI-779) — Letrozole 2.5 mg daily + Temsirolimus (CCI-779) 10 mg daily
  Arms: A
Drug: Letrozole / Temsirolimus (CCI-779) — Letrozole 2.5 mg daily + Temsirolimus (CCI-779) intermittent 30 mg daily for five days every 2 weeks
  Other Names: Letrozole / Temsirolimus(CCI-779), Torisel
  Arms: B
Drug: Letrozole — Letrozole 2.5 mg daily
  Other Names: Letrozole alone
  Arms: C

SUMMARY:
To evaluate the preliminary activity and pharmacokinetics of 2 separate doses and schedules of orally administered Temsirolimus (CCI-779) given in combination with daily letrozole, compared to letrozole alone, in the treatment of locally advanced or metastatic breast cancer in postmenopausal women. All patients must be appropriate to receive endocrine therapy as treatment for advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with histologically confirmed, measurable locally advanced disease or metastatic breast.
* Must be appropriate to receive endocrine therapy as treatment for advanced disease (chemotherapy; prior adjuvant therapy with antiestrogens other than aromatase inhibitors; prior adjuvant or first-line metastatic therapy with tamoxifen or trastuzumab, are permitted).
* Women may either present with de novo advanced or metastatic cancer, or have had tumor progression while receiving adjuvant tamoxifen or at any time after completing adjuvant tamoxifen, or have had tumor progression while receiving first-line metastatic therapy with tamoxifen.

Exclusion Criteria:

* Patients having known central nervous system (CNS) metastases.
* Prior therapy with Temsirolimus (CCI-779) or aromatase inhibitors.
* Tamoxifen, or other hormonal therapy, in the metastatic or adjuvant setting within 1 week prior to day 1 of treatment on study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2002-12; Primary Completion 2005-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066A1-204&StudyName=Study%20Evaluating%20CCI-779%20In%20Breast%20Neoplasms

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the initial protocol, doses of CCI-779 were 25 mg daily and 75 mg intermittent; per protocol amendment, dosing was modified to 10 mg daily and 30 mg intermittent. All dose levels are included in the reporting groups.
Groups:
- Let 2.5 mg Plus 10 mg Daily CCI-779: Letrozole (Let) 2.5 milligrams (mg) daily administered with a 10 mg daily dose of Temsirolimus (CCI-779).
- Let 2.5 mg Plus 30 mg Intermittent CCI-779: Letrozole (Let) 2.5 mg administered daily with a 30 mg intermittent dose (daily for 5 days every 2 weeks) of Temsirolimus (CCI-779).
- Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779: Letrozole (Let) 2.5 mg administered daily; permitted to cross-over at the time of progression to single-agent intermittent 75 mg dose (daily for 5 days every 2 weeks) of Temsirolimus (CCI-779).
- Let 2.5 mg Plus 25mg Daily CCI-779: Letrozole (Let) 2.5 mg administered daily with a 25 mg daily dose of Temsirolimus (CCI-779).
- Let 2.5 mg Plus 75 mg Intermittent CCI-779: Letrozole (Let) 2.5 mg administered daily with a 75 mg intermittent dose (daily for 5 days every 2 weeks) of Temsirolimus (CCI-779).
Period: Overall Study
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Started | 33 | 30 | 33 | 6 | 6
Completed | 0 | 0 | 3 | 1 | 0
Not Completed | 33 | 30 | 30 | 5 | 6
Not completed — Disease progression | 24 | 17 | 24 | 2 | 2
Not completed — Adverse Event | 4 | 7 | 2 | 2 | 2
Not completed — Other | 2 | 3 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 1 | 0
Not completed — Symptomatic deterioration | 1 | 1 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779 | Total
Number analyzed (Participants) | 33 | 30 | 33 | 6 | 6 | 108
Age Continuous [Mean (Standard Deviation); unit: years] | 62.21 (11.87) | 62.83 (8.39) | 60.85 (9.79) | 61.83 (9.83) | 60.00 (9.65) | 61.82 (9.98)
Sex/Gender, Customized [Number; unit: participants]
  Female | 33 | 30 | 33 | 6 | 6 | 108

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: OR measured as Complete response (CR) or Partial response (PR) confirmed by assessments performed no less than 4 weeks after the criteria for the response are first met. CR=disappearance of all target and non-target lesions with normalization of tumor marker level; PR=at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, referencing the screening sum LD. Target lesions=all measurable lesions up to 5 lesions per organ (10 lesions in total), representative of all involved organs, if possible; recorded and measured at screening. Non-target lesions=all other lesions.
Time Frame: Baseline, every 4 cycles (1 cycle is defined as a 14 day duration) up to Cycle 25, then every 6 cycles until disease progression
Population: Intent to treat population (ITT) defined as all participants randomized in the study. Final efficacy analysis was not conducted because the development of temsirolimus (CCI-779) for the treatment of breast cancer was terminated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants With Best Overall Response (Clinical Benefit)
Description: Best response (CR, PR, or stable disease (SD) lasting ≥6 months) recorded from baseline to disease progression or recurrence (Progressive disease [PD]). CR=disappearance of all target and non-target lesions with normalization of tumor marker level; PR is ≥30% decrease in sum of LD of target lesions; SD=neither sufficient shrinkage to=PR nor sufficient increase to=PD, referencing smallest sum LD since treatment started; PD is ≥20% increase in sum of LD of target lesions referencing smallest sum of LD; appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline, every 4 cycles (1 cycle is defined as a 14 day duration) up to Cycle 25, then every 6 cycles until disease progression)
Population: ITT; Final efficacy analysis was not conducted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Time to Disease Progression
Description: Number of days to disease progression defined as the interval from the date of randomization until the first date that recurrence or progression is documented; progression (at least 20% increase in the sum of the LD of target lesions taking as reference the smallest sum of LD; appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions).
Time Frame: as for outcome 2
Population: ITT; Final efficacy analysis was not conducted.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Time to Treatment Failure
Description: Number of days to treatment failure defined as interval from start of treatment to first date of progressive disease (at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD since the treatment started; appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions) or death or discontinuation of treatment due to Adverse Event, censored at last evaluation.
Time Frame: Baseline until Progressive disease, death, or discontinuation of study treatment
Population: ITT; Final efficacy analysis was not conducted.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Exhibiting Freedom From Progression
Description: Freedom from progression defined as CR (disappearance of all target and non-target lesions with normalization of tumor marker level), PR (at least a 30% decrease in sum of the LD of target lesions taking as reference the screening sum LD), or SD (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD [at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD since the treatment started; appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions]).
Time Frame: Baseline, 8 weeks, 6 months, 12 months, and 24 months
Population: ITT; Final efficacy analysis was not conducted.
Measure: Number; unit: percentage of participants
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Duration of Response
Description: Duration of response is measured from the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that reoccurrence or PD is objectively documented, taking as reference for PD the smallest measurements recorded since the treatment started. SD is measured from the start of the treatment until the criteria for disease progression are met, taking as reference the smallest measurements recorded since the treatment started; the minimal time interval for duration of SD is 8 weeks.
Time Frame: as for outcome 2
Population: ITT; Final efficacy analysis was not conducted.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Survival
Description: Number of participants with survival (alive) in the interval from start of treatment to last contact for participant or death as a result of any cause.
Time Frame: Baseline, every 4 cycles (1 cycle is defined as a 14 day duration) until death
Population: ITT; Final efficacy analysis was not conducted.
Measure: Number; unit: participants
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Health Outcomes Assessment: EuroQol (EQ-5D) Health State Profile Score
Description: EQ-5D is a self-administered questionnaire to assess health-related quality of life in 5 domains (mobility, self care, usual activities, pain or discomfort, and anxiety or depression). Scores from the 5 domains are used to calculate the Health State Profile Score as a single index value; range: 0.0 (death) to 1.0 (perfect health); higher scores indicate a better health state.
Time Frame: Prior to baseline, Cycle 7 (Week 12) and final visit (within 15 days of stopping study treatment)
Population: ITT; Final efficacy analysis was not conducted.
Measure: Number; unit: scores on a scale
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Health Outcomes Assessment: European Organization for Research and Treatment of Cancer Quality of Life Questionaire (EORTC QLQ) BR23
Description: Assess specificity of breast cancer symptoms relevant to participant's perceived quality of life (disease related symptoms of dry mouth, eye pain, hair loss, hot flushes, attractiveness, future health, sexual activity, arm or shoulder pain, breast pain, swollen breast, and skin problems on the breast). 23-item assessment of symptoms or problems during the past week (items 1-13 and 17-23) or during the past 4 weeks (items 14-16); range from 1 (not at all) to 4 (very much). Index scores transformed and range from 0 to 100; higher scores indicate higher level of functioning and quality of life.
Time Frame: Prior to baseline, Cycle 7 (Week 12) and final visit (within 15 days of stopping study treatment)
Population: ITT; Final efficacy analysis was not conducted.
Measure: Number; unit: scores on a scale
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Antitumor Response in Relation to Expression of Akt Phosphorylation, Cyclin D1, PTEN, and p27
Description: Number of participants with antitumor response (CR [disappearance of all target and non-target lesions with normalization of tumor marker level] or PR [at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, referencing the screening sum LD]) in relation to plasma levels of Akt phosphorylation, cyclin D1, PTEN, and p27.
Time Frame: Prior to baseline, after Cycle 4 (Week 8), after Cycle 8 (Week 14), and cross-over or final visit (within 15 days of stopping study treatment)
Population: ITT; Final analysis was not conducted.
Measure: Number; unit: participants
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Area Under the Concentration-time Curve (AUC) Sum
Description: Area under the concentration-time curve to infinity (AUC) measured as hours multiplied by nanograms divided by milliliters (hr*ng/mL) for CCI-779, sirolimus and letrozole. Sum is calculated as the sum of CCI-779 plus sirolimus AUCs (AUCsum).
Time Frame: Cycle 1 Day 1 (1 cycle is defined as a 14 day duration) , Cycle 3 Day 1, and Cycle 4 Day 1, Day 6, Day 9, Day 11, and Day 12
Population: ITT; Final analysis was not conducted.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: 24-hour Trough Concentration (C Trough)
Description: C trough in whole blood measured as nanograms per milliliter (ng/mL).
Time Frame: as for outcome 11
Population: ITT; Final analysis was not conducted.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone / Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Groups:
- Let 2.5 mg Alone Prior to Cross-over to 75 mg Intermit CCI-779: Letrozole (Let) 2.5 mg administered daily; permitted to cross-over at the time of progression to single-agent intermittent (intermit)75 mg dose (daily for 5 days every 2 weeks) of Temsirolimus (CCI-779). Includes events reported prior to the cross-over date for cross-over participants.
- After Cross-over to 75 mg Intermittent CCI-779: Letrozole (Let) 2.5 mg administered daily with a 25 mg daily dose of Temsirolimus (CCI-779). Includes events reported after the cross-over date for cross-over participants.
Arm/Group | Let 2.5 mg Plus 10 mg Daily CCI-779 | Let 2.5 mg Plus 30 mg Intermittent CCI-779 | Let 2.5 mg Alone Prior to Cross-over to 75 mg Intermit CCI-779 | After Cross-over to 75 mg Intermittent CCI-779 | Let 2.5 mg Plus 25mg Daily CCI-779 | Let 2.5 mg Plus 75 mg Intermittent CCI-779
Serious Adverse Events (participants affected / at risk) | 12/33 | 10/30 | 9/33 | 1/18 | 2/6 | 1/6
Other Adverse Events (participants affected / at risk) | 33/33 | 30/30 | 32/33 | 16/18 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Let 2.5 mg Plus 10 mg Daily CCI-779 (N=33) | Let 2.5 mg Plus 30 mg Intermittent CCI-779 (N=30) | Let 2.5 mg Alone Prior to Cross-over to 75 mg Intermit CCI-779 (N=33) | After Cross-over to 75 mg Intermittent CCI-779 (N=18) | Let 2.5 mg Plus 25mg Daily CCI-779 (N=6) | Let 2.5 mg Plus 75 mg Intermittent CCI-779 (N=6)
Cellulitis (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 — Organ System "General disorders" equivalent to COSTART "Body as a whole".
Death (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Infection (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Sepsis (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Accidental injury (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Organ System "Cardiac disorders" equivalent to COSTART "Cardiovascular system".
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Congestive heart failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hematoma (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hemorrhage (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolus (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 — Organ System "Gastrointestinal disorders" equivalent to COSTART "Digestive system".
Mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal carcinoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomach ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Organ System "Endocrine disorders" equivalent to COSTART "Endocrine system".
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Organ System "Blood and lymphatic system disorders" equivalent to COSTART "Hemic and lymphatic system".
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 — Organ System "Metabolism and nutrition disorders" equivalent to COSTART "Metabolic and nutritional".
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Organ System "Musculoskeletal and connective tissue disorders" equivalent to COSTART "Musculoskeletal system".
Spinal cord compression (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 — Organ System "Nervous system disorders" equivalent to COSTART "Nervous system".
Delirium (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 — Organ System "Respiratory, thoracic, and mediastinal disorders" equivalent to COSTART "Respiratory system".
Lung edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung infiltration NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Organ System "Renal and urinary disorders" equivalent to COSTART "Urogenital system".
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Reaction unevaluable (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 — Organ System "Investigations" equivalent to COSTART "Terms not classifiable".
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Let 2.5 mg Plus 10 mg Daily CCI-779 (N=33) | Let 2.5 mg Plus 30 mg Intermittent CCI-779 (N=30) | Let 2.5 mg Alone Prior to Cross-over to 75 mg Intermit CCI-779 (N=33) | After Cross-over to 75 mg Intermittent CCI-779 (N=18) | Let 2.5 mg Plus 25mg Daily CCI-779 (N=6) | Let 2.5 mg Plus 75 mg Intermittent CCI-779 (N=6)
Asthenia (General disorders) | 15 | 21 | 20 | 10 | 5 | 6
Pain (General disorders) | 12 | 12 | 12 | 4 | 1 | 1
Headache (General disorders) | 11 | 11 | 10 | 4 | 2 | 2
Back pain (General disorders) | 9 | 10 | 12 | 3 | 1 | 1
Infection (General disorders) | 9 | 8 | 9 | 1 | 3 | 2
Abdominal pain (General disorders) | 3 | 9 | 9 | 1 | 2 | 1
Chest pain (General disorders) | 6 | 4 | 3 | 1 | 0 | 1
Fever (General disorders) | 4 | 3 | 5 | 3 | 0 | 1
Accidental injury (General disorders) | 1 | 5 | 4 | 2 | 0 | 0
Flu syndrome (General disorders) | 4 | 1 | 2 | 2 | 1 | 0
Neck pain (General disorders) | 2 | 3 | 3 | 0 | 0 | 0
Cellulitis (General disorders) | 2 | 2 | 1 | 1 | 0 | 0
Chills (General disorders) | 2 | 3 | 2 | 0 | 0 | 0
Face edema (General disorders) | 4 | 2 | 1 | 3 | 0 | 0
Pelvic pain (General disorders) | 2 | 3 | 1 | 1 | 0 | 1
Lab test abnormal (General disorders) | 2 | 2 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 1 | 0 | 0 | 0 | 1
Neoplasm (General disorders) | 0 | 2 | 1 | 0 | 0 | 0
Sepsis (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Allergic reaction (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Generalized edema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Abscess (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain substernal (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Moniliasis (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Vasodilatation (Cardiac disorders) | 6 | 2 | 11 | 1 | 1 | 0
Hypertension (Cardiac disorders) | 4 | 5 | 2 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 2 | 0 | 0 | 0 | 0
Hemorrhage (Cardiac disorders) | 2 | 0 | 2 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Congestive heart failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spider vein (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiovascular physical finding (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Palpitation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Valvular heart disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Varicose vein (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 13 | 15 | 6 | 9 | 4 | 2
Mucositis (Gastrointestinal disorders) | 10 | 15 | 2 | 10 | 4 | 4
Nausea (Gastrointestinal disorders) | 7 | 11 | 10 | 5 | 2 | 3
Anorexia (Gastrointestinal disorders) | 9 | 12 | 6 | 5 | 2 | 2
Constipation (Gastrointestinal disorders) | 9 | 3 | 6 | 1 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 8 | 2 | 4 | 4 | 3
Vomiting (Gastrointestinal disorders) | 6 | 5 | 5 | 4 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 3 | 2 | 2 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 3 | 1 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 3 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0 | 2
Oral moniliasis (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1 | 0
Rectal disorder (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0 | 0
Gamma glutamyl transpeptidase increased (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0
Glossitis (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Mouth pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Stomach ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal physical finding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gum hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gum hyperplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hiatal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Periodontal abscess (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stools abnormal (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Endocrine disorders) | 1 | 2 | 0 | 1 | 0 | 0
Goiter (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 4 | 3 | 1 | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 0 | 1 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 5 | 2 | 2 | 1 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 4 | 2 | 2 | 3 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 2 | 3 | 0
Lymphedema (Blood and lymphatic system disorders) | 2 | 3 | 0 | 2 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1
Ecchymosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Granulocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral edema (Metabolism and nutrition disorders) | 16 | 11 | 5 | 4 | 4 | 2
Hyperlipemia (Metabolism and nutrition disorders) | 9 | 9 | 4 | 3 | 3 | 3
Hypercholesteremia (Metabolism and nutrition disorders) | 8 | 11 | 4 | 1 | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 10 | 2 | 2 | 0 | 1
Weight loss (Metabolism and nutrition disorders) | 8 | 5 | 1 | 2 | 1 | 1
SGOT increased (Metabolism and nutrition disorders) | 3 | 5 | 4 | 3 | 0 | 2
SGPT increased (Metabolism and nutrition disorders) | 3 | 5 | 3 | 4 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 7 | 4 | 0 | 3 | 0 | 1
Edema (Metabolism and nutrition disorders) | 5 | 3 | 1 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 1 | 1 | 1 | 2 | 0
Lactic dehydrogenase increased (Metabolism and nutrition disorders) | 4 | 1 | 3 | 1 | 0 | 1
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 2 | 3 | 3 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 1 | 0 | 0
Creatinine increased (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hyperchloremia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 0 | 0
BUN increased (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0
Bilirubinemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypoproteinemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Weight gain (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypochloremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thirst (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 13 | 12 | 5 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 7 | 7 | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 6 | 3 | 0 | 0
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 1 | 0 | 1
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal anomaly (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Bone necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myasthenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tetany (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Nervous system disorders) | 7 | 7 | 5 | 2 | 0 | 0
Depression (Nervous system disorders) | 5 | 5 | 6 | 1 | 1 | 1
Paresthesia (Nervous system disorders) | 3 | 4 | 3 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 4 | 5 | 0 | 0 | 0
Anxiety (Nervous system disorders) | 2 | 1 | 3 | 0 | 1 | 0
Vertigo (Nervous system disorders) | 2 | 1 | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 1
Hypesthesia (Nervous system disorders) | 0 | 2 | 1 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Emotional lability (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hyperesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Neuropathic pain (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abnormal gait (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hostility (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Incoordination (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Libido decreased (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
emory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nervousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Phantom pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ptosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thinking abnormal (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abnormal dreams (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stupor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 7 | 2 | 2 | 1
Cough increased (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 7 | 4 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 0 | 2 | 1 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 7 | 3 | 1 | 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 5 | 1 | 1 | 2
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 3 | 1 | 0 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 1 | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1 | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 1 | 0
Lung infiltration NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Nose dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary physical finding (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 13 | 6 | 7 | 4 | 2 — Organ System "Skin and subcutaneous tissue disorders" equivalent to COSTART "Skin and appendages".
Nail disorder (Skin and subcutaneous tissue disorders) | 10 | 9 | 0 | 3 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 7 | 0 | 5 | 2 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 4 | 6 | 1 | 1 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 3 | 7 | 1 | 4 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 5 | 3 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4 | 2 | 3 | 2 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 3 | 0 | 0
Fungal dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 1
Maculopapular rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 2 | 0 | 0
Sweating (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 0 | 0 | 0
Exfoliative dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 1 | 0
Folliculitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1
Herpes simplex (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 4 | 0 | 0
Pruritic rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0
Skin discoloration (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1 | 0
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pustular rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Vesiculobullous rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Melanosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 5 | 3 | 2 | 3 | 1 | 0 — Organ System "Eye disorders" equivalent to COSTART "Special senses".
Abnormal vision (Eye disorders) | 1 | 3 | 1 | 0 | 1 | 0
Eye disorder (Eye disorders) | 2 | 2 | 1 | 0 | 0 | 1
Dry eyes (Eye disorders) | 1 | 2 | 0 | 1 | 2 | 0
Cataract specified (Eye disorders) | 0 | 3 | 0 | 1 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 2 | 1 | 0 | 0 — Organ System "Ear and labyrinth disorders" equivalent to COSTART "Special senses".
Ear disorder (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0
Otitis externa (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 3 | 3 | 1 | 5 | 2 | 1
Dysuria (Renal and urinary disorders) | 3 | 2 | 2 | 1 | 1 | 1
Cystitis (Renal and urinary disorders) | 3 | 2 | 0 | 0 | 1 | 0
Vaginal moniliasis (Renal and urinary disorders) | 4 | 1 | 0 | 1 | 0 | 0
Vaginal dryness (Renal and urinary disorders) | 2 | 1 | 1 | 1 | 0 | 0
Metrorrhagia (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0
Vaginal hemorrhage (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0
Breast pain (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Leukorrhea (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginitis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Reaction unevaluable (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 — Organ System "Investigations" equivalent to COSTART "Terms not classifiable".
Local reaction to procedure (Investigations) | 1 | 2 | 1 | 2 | 0 | 0 — Organ System "Investigations" equivalent to COSTART "Adverse event associated with miscellaneous factors".
Allergic reaction other than drug (Investigations) | 2 | 1 | 0 | 0 | 0 | 0
Laboratory events not classified (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Taste loss (Nervous system disorders) | 3 | 0 | 1 | 2 | 2 | 2
Taste perversion (Nervous system disorders) | 0 | 2 | 0 | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
Clinical development of oral temsirolimus for treatment of locally advanced or metastatic breast cancer was terminated by Wyeth based on the results of a phase 3 clinical study with the combination temsirolimus and letrozole.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.